CLINICAL TRIAL: NCT02618668
Title: Haemodynamic Stability of Ketamine / Propofol Admixture "Ketofol" in Patient Undergoing Endoscopic Retrograde Cholangio Pancreatography
Brief Title: Haemodynamic Stability of Ketamine/Propofol Admixture "Ketofol" in Patient Undergoing Endoscopic Retrograde Cholangio Pancreatography
Acronym: Assiutu
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, m mostfa youssef mekky, resident of anesthesia and ICU, Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Momen01098983009
Record Dates: First submitted 2015-11-16; First posted 2015-12-01 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Pancreatitis; Cholangitis
MeSH Terms: conditions — Pancreatitis; Cholangitis | interventions — Ketamine; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Ketamine / Propofol Admixture (Experimental): Ketamine / Propofol Admixture: I.V propofol-ketamine 3:1 mixture(%1 15 ml propofol + 1 ml 50mg/ml ketamine+ 4 ml saline in a 20-ml syringe which resulted in 0.25 mg.ml-1 ketamine and 0.75 mg.ml-1 propofol.
  Interventions: Drug: Ketamine / Propofol Admixture
- Propofol (Active Comparator): I.V propofol 2 mg/kg
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Ketamine / Propofol Admixture — propofol-ketamine 3:1 mixture(%1 15 ml propofol + 1 ml 50mg/ml ketamine+4 ml saline in a 20-ml syringe which resulted in0.25 mg.ml-1 ketamine and 0.75 mg.ml-1 propofol
  Arms: Ketamine / Propofol Admixture
Drug: Propofol — 2 mg/kg I.V
  Arms: Propofol

SUMMARY:
The investigators aim to evaluate the effect of Ketamine/Propofol Admixture on hemodynamic stability, recovery time ,patient & doctor satisfaction scores during Endoscopic Retrograde Cholangiopancreatography.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists ( I ,II )

Exclusion Criteria:

1. Presence of liver and/or kidney failure, neuropsychiatric disorders, morbid obesity.
2. History of substance abuse or dependence.
3. History of serious adverse effects related to anesthetics (e.g. allergic reactions), a family history of reactions to the study drugs.
4. Pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2015-07; Primary Completion 2018-07 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
mean arterial blood pressure from baseline of patient undergoing Endoscopic Retrograde Cholangio pancreatography | every 5 minutes up to 30minutes
saturation of oxygen from baseline of undergoing Endoscopic Retrograde Cholangio pancreatography | every 5 minutes up to 30 minutes
Heart rate( beat/minute) from baseline of patient | every 5 minutes up to 30 minutes
Recovery score of patient | up to 10 minutes after the end of procedure

SECONDARY OUTCOMES:
patient and doctor satisfaction score | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed A Bakr, Prof., Study Chair — Assiut University; Nagwa m osman, Asst.prof., Study Director — Assiut University
Locations (1):
- Assiut university hospital, Asyut, Egypt